CLINICAL TRIAL: NCT02976584
Title: Incidence of Epileptic Potentials During Cardiac Surgery and Postoperative Neurological Outcome: A Prospective Observational Study
Brief Title: Epileptic Potentials During Cardiac Surgery and Association With Postoperative Neurological Outcome
Acronym: EPOCAS
Status: Completed | Type: Observational
Sponsor: Heiko Kaiser (Other)
Responsible Party: Sponsor-Investigator, Heiko Kaiser, Dr. med., Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Other Study IDs: KEK210/15
Record Dates: First submitted 2016-10-19; First posted 2016-11-29 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Epilepsy; Cardiac Disease; Peroperative Complications; Anesthesia; Adverse Effect; Ischemia, Cerebral
Keywords: EEG; Cardiac Surgery; Seizure; Tranexamic acid
MeSH Terms: conditions — Epilepsy; Heart Diseases; Intraoperative Complications; Brain Ischemia; Seizures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Primarily, the investigators want to test the hypothesis that it is possible to detect epileptiform EEG during cardiac surgery under general anesthesia.

Furthermore, the investigators will examine if those epileptic potentials coincide, follow or are unrelated to ischemic events detected by EEG or Near-infrared spectroscopy (NIRS). Finally, the investigators will look for independent associations between intraoperative seizures (with or without ischemic events) and postoperative neurological outcome, as well as between intraoperative seizures (with or without ischemic events) and the total amount of TXA given.

DETAILED DESCRIPTION:
The investigators will follow the STROBE guidelines to perform this prospective observational study. All patient demographics, co-morbidities and surgical details that are relevant to calculate the EuroSCORE will be recorded using our institutional automatic anesthesia record system. Laboratory tests will be performed according to our clinical standard before cardiac surgery. General anesthesia and surgery will be performed according to attending physician's preferences. Invasive arterial blood pressure, central line and transesophageal echocardiography (TEE) are all standard procedures. Before induction of anesthesia a two channel EEG will be installed on the forehead with reference electrode on FPZ, other electrodes on A1-F3 & A2-F4. A Narcotrend Compact M Monitor will be connected to evaluate depth of anesthesia continuously during the operation, but also automatically stores EEG data (with a rate of 128Hz) to screen for epileptic activity or/and ischemic episodes. This monitor is standard practice in our cardiovascular division.

Patients at higher risk for intraoperative cerebral ischemic events (stenosis of carotid artery, deep hypothermic cardiac arrest, history of stroke/prind/TIA, severe aortic atherosclerotic disease) do receive bilateral frontal brain oxygenation/perfusion monitoring with Near-infrared spectroscopy (NIRS) as part of standard practice at our institution. After the administration of the anticoagulant heparin for cardiopulmonary bypass, tranexamic acid is given intravenously as our clinical standard according to the BART trial. All other intraoperative administrations of drugs, blood transfusions and hemodynamic management will be according to the responsible cardiac anesthesiologist and cardiac surgeon. Following surgery patients will be transported to the ICU under deep sedation according to the anesthesia team. As standard operation procedure the responsible ICU attending or resident is evaluating cardiac surgery patients every hours while intubated and at least twice per shift if awake (4 times per day) for neurological deficits. A neurological deficit is defined as patient developing a new onset motor, sensory, or cognitive dysfunction (e.g., hemiplegia, hemiparesis, aphasia, sensory deficit, impaired memory) that persists for 24 or more hours due to embolic, thrombotic, or hemorrhagic vascular accident or stroke. Special trained ICU nurses evaluate the Richmond Agitation Sedation Scale (RASS) on an hourly basis. The time from stopping sedation until reaching a RASS of zero will be used to determine (delayed) time to awakening. The appropriateness of timing to stop the sedation is up to the treating ICU team.

Standard practice is, that cardiac enzymes are measured all 6 hours for the first 48 hours, according to clinical judgement thereafter, but at least once daily until discharge from the ICU. New myocardial infarction will be defined as Troponin values >10x99th percentile URL during the first 48 h following cardiac surgery, occurring from a normal baseline Troponin value (≤99th percentile URL). In addition, either (i) new pathological Q waves or new LBBB, or (ii) angiographically documented new graft or new native coronary artery occlusion, or (iii) imaging evidence of new loss of viable myocardium or new regional wall motion abnormality.

Pulmonary and respiratory complications will be noted as (1) pneumonia, (2) prolonged intubation of > 24 hours, (3) re-intubation, (4) TRALI or ARDS, as well as (5) tracheostomy due to weaning failure.

Renal complication is defined as acute renal failure (ARF) requiring dialysis during the postoperative period. The indication for dialysis include uremia, volume overload, or biochemical abnormalities and are based on clinical judgment of the treating ICU team.

The exact time on the ICU and on the ventilator is automatically recorded in the patient data management system (PDMS) and will be recorded on the day of ICU discharge and/or extubation. All postoperative diagnosis of complications will be gathered from the involved intensivist, cardiac surgeon, cardiologist, neurologist, radiologist and other consulted specialists. Mortality will be evaluated for in hospital only.

The postoperative course of all included patients will be followed until discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are undergoing elective or emergent cardiac or major aortic surgery with cardiopulmonary bypass.

Exclusion Criteria:

* Patients refusing to consent to our institutional protected health information policy on the consent document for anesthesia or the general consent of the INSELSPITAL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are undergoing elective or emergent cardiac or major aortic surgery with cardiopulmonary bypass and are at least 18 years old.
  Single-centre: INSELSPITAL, Bern, Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 1067 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2017-11-24 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Incidence of intraoperative epileptic seizures | Up to 1 day

SECONDARY OUTCOMES:
Neurologic injury (Stroke, PRIND, TIA) | up to 30 days
Delayed wakening from anesthesia | up to 30 days
Postoperative cardiac/pulmonary/renal complications | up to 30 days
Mortality | up to 30 days
Time on the ventilator | up to 30 days
ICU length of stay | up to 30 days
Hospital length of stay | up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Kaiser, MD, Principal Investigator — Dept. of Anesthesiology and Pain Therapy, Division of Cardiovascular Anesthesia, University Hospital Inselspital, Berne
Locations (1):
- University Hospital Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ebensperger M, Kreuzer M, Kratzer S, Hight D, Kaiser HA, Schneider G, Schwerin S. Evaluating the performance of the NarcotrendR EEG index during anaesthesia for cardiothoracic surgery: a single-centre retrospective study. BMC Anesthesiol. 2025 Nov 14;25(1):559. doi: 10.1186/s12871-025-03500-5. PMID 41239249
- [Derived] Hight D, Ehrhardt A, Lersch F, Luedi MM, Stuber F, Kaiser HA. Lower alpha frequency of intraoperative frontal EEG is associated with postoperative delirium: A secondary propensity-matched analysis. J Clin Anesth. 2024 May;93:111343. doi: 10.1016/j.jclinane.2023.111343. Epub 2023 Nov 22. PMID 37995609
- [Derived] Hight D, Schanderhazi C, Huber M, Stuber F, Kaiser HA. Age, minimum alveolar concentration and choice of depth of sedation monitor: examining the paradox of age when using the Narcotrend monitor: A secondary analysis of an observational study. Eur J Anaesthesiol. 2022 Apr 1;39(4):305-314. doi: 10.1097/EJA.0000000000001576. PMID 34313611
- [Derived] Kaiser HA, Hirschi T, Sleigh C, Reineke D, Hartwich V, Stucki M, Rummel C, Sleigh J, Hight D. Comorbidity-dependent changes in alpha and broadband electroencephalogram power during general anaesthesia for cardiac surgery. Br J Anaesth. 2020 Oct;125(4):456-465. doi: 10.1016/j.bja.2020.06.054. Epub 2020 Jul 31. PMID 32747077
- [Derived] Kaiser HA, Peus M, Luedi MM, Lersch F, Krejci V, Reineke D, Sleigh J, Hight D. Frontal electroencephalogram reveals emergence-like brain activity occurring during transition periods in cardiac surgery. Br J Anaesth. 2020 Sep;125(3):291-297. doi: 10.1016/j.bja.2020.05.064. Epub 2020 Jul 15. PMID 32682555
- See also: Ordinance on Human Research with the Exception of Clinical Trials (Human Research Ordinance, HRO) — http://www.admin.ch/opc/en/classified-compilation/20121177/index.html